CLINICAL TRIAL: NCT00483951
Title: Suburban/NHLBI Cardiovascular Disease Screening Protocol
Brief Title: Cardiovascular Disease Screening
Status: Terminated | Type: Observational
Why Stopped: Per IRB recommendation, a separate protocol will be prepared for retrospective data analysis. The current protocol does not have specific hypotheses.
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070157; 07-H-0157
Record Dates: First submitted 2007-06-07; First posted 2007-06-08 (Estimated); Last update posted 2021-07-29 (Actual); Status verified 2020-11

CONDITIONS: Congenital Heart Disease; Atherosclerosis; Myocardial Ischemia; Myocardial Infarction; Acquired Heart Disease
Keywords: Transthoracic echocardiography; Ischemia; Cardiovascular Disease
MeSH Terms: conditions — Heart Defects, Congenital; Atherosclerosis; Myocardial Ischemia; Myocardial Infarction; Ischemia; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Patients with known or suspected cardiovascular disease: Patients referred to protocol with known or suspected cardiovascular disease for further evaluation.
  Interventions: Device: Toshiba Aquilion ONE CT; Device: SWiemens MRI scanner

INTERVENTIONS:
Device: Toshiba Aquilion ONE CT — The Toshiba Aquilion ONE CT system has the ability to acquire whole organ volume images in a single rotation by utilizing an x-ray detector that is configured as 320 detector rows with a 0.5 mm width, providing a z-axis coverage of 16 cm of anatomy.
Device: SWiemens MRI scanner — Investigational or research MRI coils may be used in the protocol. The coils are noninvasive devices external to the body. The coils act as antennae to receive small radiofrequency signals out of the body. Coils of the type we use are used daily in clinical MRI practice.

SUMMARY:
This study will evaluate volunteers 18 years of age and older to see if they qualify for one of NHLBI s research studies. Tests include the following:

* General medical evaluation, which may include blood tests, chest x-ray, electrocardiogram (ECG) and echocardiogram (heart ultrasound).
* Other tests as appropriate, such as magnetic resonance imaging (MRI), cardiac computed tomography (CT scan of the heart), nuclear stress test and echocardiography stress test.
* X-ray contrast studies of the heart and blood vessels. (These may be excluded in patients with kidney risk factors.)

DETAILED DESCRIPTION:
This is a screening protocol. This protocol allows two functions: 1) the protocol allows physicians in the Suburban/NHLBI Cardiovascular Imaging program to evaluate patients referred to the program with clinically indicated studies and research studies. 2) It is also designed to determine if patients may be suitable candidates for one of our NHLBI research protocols.

Patients greater than or equal to 18 years of age referred for possible cardiovascular disease will be enrolled in the protocol for a period of one year. At one year, patients will either be: 1) transferred to one of our specific research MRI or CT protocols, 2) removed from the screening protocol and made inactive, or 3) re-enrolled on the screening protocol with the patient s consent.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

No one will be excluded from this study based on race, gender, or ethnicity.

A. General Inclusion Criteria:

* Age greater than or equal to 18
* Capable of giving informed consent.

B. General Exclusion Criteria:

* Pregnant women (uncertain patients will have urine or blood testing).
* Decompensated heart failure (unable to lie flat in bed).

Test Specific Exclusion Criteria:

A. CT Exclusion Criteria (excludes contrast enhanced CT scan only):

* Allergy to iodinated contrast agent excludes contrast enhanced CT research studies.
* Multiple myeloma.
* Patients with severe kidney disease (eGFR less than 30 mL/min/1.73 m(2).

B. Beta Antagonist Exclusions (excluded the use of beta blocker only):

* Asthma or severe chronic lung disease/emphysema with regular use of inhaler.
* Decompensated heart failure.

C. MRI Exclusion Criteria (excludes MRI scan only):

* Cardiac pacemaker or implantable defibrillator.
* Cerebral aneurysm clip.
* Neural stimulator (e.g. TENS-Unit).
* Any type of ear implant.
* Metal in eye (e.g. from machining).
* Any implanted device (e.g. insulin pump, drug infusion device).

D. Exclusions from MRI contrast agents:

* Lactating women unless they are willing to discard breast milk for 24 hours.
* Severe kidney disease (less than 30 mL/min/1.73 m(2).

E. Vasodilator Exclusions (excludes some vasodilator stress testing):

* Asthma or chronic obstructive pulmonary disease (emphysema) actively treated with bronchodilators or leukotriene receptor antagonists (albuterol, seravent, atrovent, montelukast singulair, zafirlukast Accolate. These conditions only exclude adenosine and dipyridamole.
* Second degree (Type II) and third degree atrioventricular heart block.

F. Exclusions from Dobutamine stress MRI only:

* Severe problems with heart rhythms.
* Severe high blood pressure.

G. Exclusion criteria for atropine (given during dobutamine stress echocardiography when target heart rate not achievable with dobutamine alone).

* Narrow angle glaucoma.
* Known or suspected severe bladder outlet obstruction due to prostatic hypertrophy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients > 18 years of age referred for possible cardiovascular disease will be enrolled in the protocol for a period of one year.
  At one year, patients will either be: 1) transferred to one of our specific research MRI or CT protocols, 2) removed from the screening protocol and made inactive, or 3) re-enrolled on the screening protocol with the patient's consent.
Sampling Method: Non-Probability Sample
Enrollment: 1325 (Actual)
Dates: Start 2008-01-28 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2020-11-03 (Actual)

PRIMARY OUTCOMES:
Complete characterization of patients for screening purpose onto a research protocol. | Ongoing
  Complete characterization of patients for the purpose of deciding whether they are eligible for research protocols run by the Cardiovascular Branch.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew E Arai, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (2):
- United States (2):
  - Suburban Hospital, Bethesda, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Escolar E, Weigold G, Fuisz A, Weissman NJ. New imaging techniques for diagnosing coronary artery disease. CMAJ. 2006 Feb 14;174(4):487-95. doi: 10.1503/cmaj.050925. PMID 16477061
- [Background] White CS, Kuo D, Kelemen M, Jain V, Musk A, Zaidi E, Read K, Sliker C, Prasad R. Chest pain evaluation in the emergency department: can MDCT provide a comprehensive evaluation? AJR Am J Roentgenol. 2005 Aug;185(2):533-40. doi: 10.2214/ajr.185.2.01850533. PMID 16037533
- [Background] Hendel RC, Patel MR, Kramer CM, Poon M, Hendel RC, Carr JC, Gerstad NA, Gillam LD, Hodgson JM, Kim RJ, Kramer CM, Lesser JR, Martin ET, Messer JV, Redberg RF, Rubin GD, Rumsfeld JS, Taylor AJ, Weigold WG, Woodard PK, Brindis RG, Hendel RC, Douglas PS, Peterson ED, Wolk MJ, Allen JM, Patel MR; American College of Cardiology Foundation Quality Strategic Directions Committee Appropriateness Criteria Working Group; American College of Radiology; Society of Cardiovascular Computed Tomography; Society for Cardiovascular Magnetic Resonance; American Society of Nuclear Cardiology; North American Society for Cardiac Imaging; Society for Cardiovascular Angiography and Interventions; Society of Interventional Radiology. ACCF/ACR/SCCT/SCMR/ASNC/NASCI/SCAI/SIR 2006 appropriateness criteria for cardiac computed tomography and cardiac magnetic resonance imaging: a report of the American College of Cardiology Foundation Quality Strategic Directions Committee Appropriateness Criteria Working Group, American College of Radiology, Society of Cardiovascular Computed Tomography, Society for Cardiovascular Magnetic Resonance, American Society of Nuclear Cardiology, North American Society for Cardiac Imaging, Society for Cardiovascular Angiography and Interventions, and Society of Interventional Radiology. J Am Coll Cardiol. 2006 Oct 3;48(7):1475-97. doi: 10.1016/j.jacc.2006.07.003. No abstract available. PMID 17010819
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2007-H-0157.html